CLINICAL TRIAL: NCT01694121
Title: Evaluating a Structural and Behavioral HIV Risk Reduction Program for Black Men
Acronym: MENCount
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Anita Raj, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH096657 (NIH)
Record Dates: First submitted 2012-09-22; First posted 2012-09-26 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: HIV
Keywords: HIV prevention; African American men; evaluation study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEN Count (Experimental): 3 session HIV intervention including a) HIV risk reduction, inclusive of gender equity and healthy relationship counseling and b) case management support for stable employment and housing.
  Interventions: Behavioral: MEN Count
- Comparison (Active Comparator): An attention comparison program similar to the MEN Count intervention in structure (3 one-on-one sessions delivered over 60-90 days) but focused on stress reduction and healthy lifestyle.
  Interventions: Behavioral: Comparison

INTERVENTIONS:
Behavioral: MEN Count — The MEN Count model integrates HIV risk reduction and gender-equity counseling with housing and employment case management via multiple one-on-one sessions delivered by a peer case manager over 60-90 day period.
  Arms: MEN Count
Behavioral: Comparison — general health intervention for men, not inclusive of HIV or relationship health
  Arms: Comparison

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Making Employment Needs (MEN) Count intervention, an HIV intervention and prevention program for heterosexual Black men. The MEN Count model integrates HIV risk reduction and gender-equity counseling with housing and employment case management via multiple one-on-one sessions delivered by a peer case manager over 60-90 day period. MEN Count was developed and pilot tested using a Community-based participatory research (CBPR) approach via funding from a National Institutes of Health (NIH) R21, in Boston, Massachusetts. A more larger scale, two-armed quasi-experimental controlled trial design will be used to test MEN Count among Black men recruited/enrolled from an STD clinic and other community-recruitment methods in Washington, DC. Study participants (N=504) will be Black men reporting heterosexual risk for HIV [unprotected sex with a woman and 2+ female sex partners in the past 6 months] and either current unemployment or homeless in the past 6 months. To evaluate the effectiveness of MEN Count, a two-armed quasi-experimental design will be conducted in which participants will receive either MEN Count or an attention comparison program similar to MEN Count in structure. We will assess program impact on reduction in number of unprotected sex episodes and incident cases of STI (Chlamydia, gonorrhea, syphilis) via survey and STI testing, respectively, at baseline and 6 and 12 month follow-ups. Additionally, quality assurance and process evaluation efforts will be conducted to ensure high quality program adherence and delivery, as well as to support program replication should the model prove effective.

ELIGIBILITY:
Inclusion Criteria: Black men aged 18 and older, reporting heterosexual risk for HIV [unprotected sex with a woman and 2+ female sex partners in the past 6 months] and either current unemployment or homeless in the past 6 months.

Exclusion Criteria: planned to leave Washington D.C., Maryland, or Virginia in the next 6 months, were cognitively impaired (based on Folstein Mini-Mental Exam at recruitment or baseline testing), and/or had self-reported health status that prohibited them from participating in the program

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 455 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Raj, PhD, Principal Investigator — UCSD; Lisa Bowleg, PhD, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: one individual was enrolled and surveyed twice. He remained in the study, but the initial survey was not included.
Period: Overall Study
Arm/Group | MEN Count | Comparison
Started | 228 | 227
Completed | 227 | 227
Not Completed | 1 | 0
Not completed — Participant used false ID, was withdrawn | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEN Count | Comparison | Total
Number analyzed (Participants) | 227 | 227 | 454
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 227 | 227 | 454
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 227 | 227 | 454
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 227 | 227 | 454
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 227 | 227 | 454
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 227 | 227 | 454
full time employment status [Count of Participants; unit: Participants] | 19 | 34 | 53
non-Viral STI [Count of Participants; unit: Participants] | 55 | 51 | 106
homeless in a shelter or on the streets in past 90 days [Count of Participants; unit: Participants] | 116 | 104 | 220

OUTCOME MEASURES:

1. Primary Outcome: Condom Use/Unprotected Sex - Redefined as Sexual Risk - 12 Month Follow-up
Description: Behavioral assessment of the ratio of protected to total number of sex episodes -- changed to sexual risk inclusive of inconsistent condom use in past 90 days + multiple sex partners + sex trade involvement. Very low sexual risk was defined as having one partner and consistent condom use. Low sexual risk was defined as having multiple partners and consistent condom use OR one partner and no/inconsistent condom use. Medium sexual risk was defined as having multiple partners, no/inconsistent condom use and not participating in transactional sex. High risk was defined as having multiple partners, no/inconsistent condom use, and participating in transactional sex. Participants reporting sex with men in the prior 90 days or who reported that they themselves or (one of) their partner(s) was HIV-positive were excluded from the sexual risk outcome given the known differential HIV risk profile for these subpopulations and small numbers of participants in each.
Time Frame: 12 month follow-up
Population: Those retained at 12 mo follow up
Measure: Count of Participants; unit: Participants
Arm/Group | MEN Count | Comparison
Number analyzed (Participants) | 120 | 123
Participants
  Very low risk | 28 | 18
  Low risk | 26 | 40
  Medium risk | 30 | 34
  High risk | 7 | 9
  Excluded or missing risk | 29 | 22

2. Secondary Outcome: Non-viral STI - 12 Month Follow-up
Description: HIV and STI testing via blood and urine tests was conducted; outcome based on non-viral STI to allow for incidence assessment and change over time
Time Frame: 12 month follow-up
Population: Participants retained at 12mo follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | MEN Count | Comparison
Number analyzed (Participants) | 120 | 123
Participants
  Positive for non-viral STI at 12mo follow-up | 17 | 15
  Negative for all non-viral STI at 12mo follow-up | 87 | 98
  Did not complete STI testing at 12mo follow-up | 16 | 10

3. Secondary Outcome: Non-viral STI - 6 Month Follow-up
Description: as for outcome 2
Time Frame: 6 month follow-up
Population: Participants retained at 6mo follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | MEN Count | Comparison
Number analyzed (Participants) | 95 | 105
Participants
  Positive for non-viral STI at 6mo follow-up | 7 | 13
  Negative for all non-viral STI at 6mo follow-up | 83 | 85
  Did not complete STI testing at 6mo follow-up | 5 | 7

4. Primary Outcome: Condom Use/Unprotected Sex - Redefined as Sexual Risk - 6 Month Follow-up
Description: as for outcome 1
Time Frame: 6 month follow-up
Population: Those retained at 6 mo follow up
Measure: Count of Participants; unit: Participants
Arm/Group | MEN Count | Comparison
Number analyzed (Participants) | 95 | 105
Participants
  Very low risk | 15 | 18
  Low risk | 32 | 29
  Medium risk | 25 | 28
  High risk | 6 | 8
  Excluded or missing risk | 17 | 22

ADVERSE EVENTS:
Time Frame: Duration of the study (up to 12 months)
Arm/Group | MEN Count | Comparison
All-Cause Mortality (participants affected / at risk) | 1/227 | 1/227
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/227
Other Adverse Events (participants affected / at risk) | 0/227 | 0/227

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT01694121/Prot_SAP_000.pdf
  • Informed Consent Form (2015-02-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT01694121/ICF_001.pdf